CLINICAL TRIAL: NCT00001629
Title: The Role of Angiotensin Type I Receptor in the Regulation of Human Coronary Vascular Function
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 970142; 97-H-0142
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-06

CONDITIONS: Atherosclerosis; Heart Failure, Congestive; Hypertension; Myocardial Infarction
Keywords: Angiotensin AT-1 Receptor; Angiotensin Receptor Antagonist; Atherosclerosis; Blood Flow; Cold Pressor Test; Endothelium; Exercise; Coronary Artery Disease; Heart Failure
MeSH Terms: conditions — Atherosclerosis; Heart Failure; Hypertension; Myocardial Infarction; Motor Activity; Coronary Artery Disease | interventions — Angiotensin II Type 1 Receptor Blockers

INTERVENTIONS:
Drug: Angiotensin II type 1 receptor antagonists

SUMMARY:
The renin angiotensin system (RAS) plays an important physiological and pathophysiological role in the control of blood pressure and plasma volume. Inhibition of the RAS is useful in the treatment of hypertension, cardiac failure and in some patients with myocardial infarction. Several recent clinical trials with angiotensin converting enzyme inhibitors (ACEI) have shown that they also reduce the incidence of myocardial infarction, but the mechanisms underlying this anti-ischemic effect are poorly understood. ACEI reduce angiotensin II synthesis and prevent bradykinin degradation. Results from ongoing studies in the Cardiology Branch (Protocol 95-H-0099) designed to investigate the link between ACEI and the vascular endothelium indicate that ACEI improve both endothelial dysfunction and metabolic coronary vasodilation, an effect that is partially mediated by bradykinin. The current protocol is designed to investigate whether the beneficial effects of ACEI on endothelial function are also partly due to inhibition of angiotensin II. The recent development of selective angiotensin II type 1 (AT1) receptor antagonists allows us to specifically examine the effects of angiotensin II on vasomotor activity.

DETAILED DESCRIPTION:
The renin angiotensin system (RAS) plays an important physiological and pathophysiological role in the control of blood pressure and plasma volume. Inhibition of the RAS is useful in the treatment of hypertension, cardiac failure and in some patients with myocardial infarction. Several recent clinical trials with angiotensin converting enzyme inhibitors (ACEI) have shown that they also reduce the incidence of myocardial infarction, but the mechanisms underlying this anti-ischemic effect are poorly understood. ACEI reduce angiotensin II synthesis and prevent bradykinin degradation. Results from ongoing studies in the Cardiology Branch (Protocol 95-H-0099) designed to investigate the link between ACEI and the vascular endothelium indicate that ACEI improve both endothelial dysfunction and metabolic coronary vasodilation, an effect that is partially mediated by bradykinin. The current protocol is designed to investigate whether the beneficial effects of ACEI on endothelial function are also partly due to inhibition of angiotensin II. The recent development of selective angiotensin II type 1 (AT1) receptor antagonists allows us to specifically examine the effects of angiotensin II on vasomotor activity.

ELIGIBILITY:
Patient must be over 18 years of age requiring diagnostic cardiac catheterization will participate.

Women on chronic estrogen therapy are eligible for the study.

Patients investigated for chest pain syndrome with normal coronary arteries with and without risk factors for atherosclerosis, patients with coronary artery disease, and patients with heart failure.

No patients with unstable angina; significant left main disease (greater than 50% stenosis); Recent myocardial infarction (less than 1 month); Pregnancy, lactation; Allergy to losartan; Renal failure (creatinine greater than 2.5 mg/dl); Inability to withdraw ACE inhibitors.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49
Dates: Start 1997-07; Study Completion 2000-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Cockcroft JR, Sciberras DG, Goldberg MR, Ritter JM. Comparison of angiotensin-converting enzyme inhibition with angiotensin II receptor antagonism in the human forearm. J Cardiovasc Pharmacol. 1993 Oct;22(4):579-84. doi: 10.1097/00005344-199310000-00011. PMID 7505360
- [Background] Goldberg MR, Tanaka W, Barchowsky A, Bradstreet TE, McCrea J, Lo MW, McWilliams EJ Jr, Bjornsson TD. Effects of losartan on blood pressure, plasma renin activity, and angiotensin II in volunteers. Hypertension. 1993 May;21(5):704-13. doi: 10.1161/01.hyp.21.5.704. PMID 8491505
- [Background] Sudhir K, MacGregor JS, Gupta M, Barbant SD, Redberg R, Yock PG, Chatterjee K. Effect of selective angiotensin II receptor antagonism and angiotensin converting enzyme inhibition on the coronary vasculature in vivo. Intravascular two-dimensional and Doppler ultrasound studies. Circulation. 1993 Mar;87(3):931-8. doi: 10.1161/01.cir.87.3.931. PMID 8383016